CLINICAL TRIAL: NCT06144775
Title: Manual Motor Planning Deficits and Performance Differences in Children With Autism Spectrum Condition: a Kinematic Analysis to Extract Objective Markers of Motor Atypia
Brief Title: A Kinematic Analysis of Motor Planning and Movement Execution of Children With Autism Spectrum Condition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2023-004
Record Dates: First submitted 2023-11-07; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism spectrum condition; motor planning; kinematic analysis; children
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with autism spectrum condition: Thirty ASC children with medium-high functioning, aged 7 to 13 years, IQ > 80, in the absence of motor deficits due to another clinical condition.
  Interventions: Other: Kinematics measures
- Children with typical development: Thirty TD children, aged 7 to 13 years, IQ > 80, in the absence of motor deficits due to clinical condition.
  Interventions: Other: Kinematics measures

INTERVENTIONS:
Other: Kinematics measures — In a single session each child will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed. The study involves the use of three blocks of tasks of the neuropsychological battery (NEPSY-II): Finger Tapping, Visuo-Motor Precision, and Manual Motor Sequences. The order within each block will be randomized.

SUMMARY:
Autism Spectrum Condition (ASC) is a behavioral syndrome characterized by a severe organizational disorder of thinking and major functions that regulate human adaptation. It is to be considered as a functional disorder, or of executive functions, whose dysfunction is expressed in the difficulty of making voluntary movements, sequentially coordinated with each other according to a purpose, and of initiating an action, planning and monitoring it by inhibiting inappropriate responses such as gesture perseveration. Literature studies suggest that, compared to children with typical development (TD) and regardless of cognitive status, children with ASC have pervasive motor dysfunction that results in universal difficulties in several aspects of motor function, including - (1) fine motricity, (2) some aspects of praxis while performing tasks based on imitation of sequences, (3) simultaneous coordination of both sides of the body during rhythmic tasks of the upper limbs, and́ (4) interpersonal coordination and synchrony. The hypothesis of the study is that by comparing these aspects in 2 groups of children with ASC and children with TD using A.I. systems, it will be possible to extract objective markers of motor deficits found in autism, facilitating the validation of measurements acquired with clinical scales. The objective of the study is to investigate the characteristics of manual motor planning and performance difficulties in children with ASC using kinematic measurements. 30 ASC children with medium-high functioning and 30 TD children, aged 7 to 13 years, IQ > 80, in the absence of motor deficits due to another clinical condition, will be recruited. The protocol will take place in a single session during which children will be video-recorded performing simple and complex rhythmic upper limb actions with a social partner. The presence of characteristic fine motor behaviors, practice errors, perseverations, movement variability, and interpersonal synchrony will be observed. The study will involve the use of 3 tasks contained in NEPSY-II: Finger tapping, Visual-motor precision, and Imitation of manual motor sequences. The videos will be recorded simultaneously and the different angles will allow hand kinematics to be extracted and analyzed with A.I. algorithms to measure displacement, velocity, acceleration, frequency and any other kinematic parameters highlighted. Thus, it is expected to identify objective markers of motor deficits found in children with ASC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism
* QI ≥ 80.

Exclusion Criteria:

* Motor deficits due to another clinical condition

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thirty children with ASD and 30 typically developing (TD) children will participate in the study. The children with ASD will be recruited and tested at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina. To be included in the study the child needs to have an ASD diagnosis based on the DSM-5 criteria from a licensed clinical child neuropsychiatrist but no established intellectual disability (ID) diagnosis. The TD children will recruit through advertisements in schools located close to the Institute. Informed consent will obtain from all subjects involved in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Reaction time and latency | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the movement's reaction time and latency in seconds (s).
Speed | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the movement's speed in millimeter per second (mm/s).
Quantity of motion | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the quantity of motion.
Frequency | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the frequency in Hertz (Hz) of the movements.
Acceleration | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the movement's acceleration in millimeter per square second (mm/s2).
Angular speed | The recording session needs approximately 20 minutes to complete.
  In a single session the children will be video-recorded while performing simple and complex rhythmic actions of the upper limbs with a social partner. The presence of characteristic motor behaviors, practice errors, perseverations, and movement variability will be observed.
  During the execution of the three blocks of tasks (finger tapping, visuo-motor precision, and manual motor sequences) four GOPRO cameras, mounted on tripods in different angles of the room, record videos simultaneously.
  The videos will be analyzed through Artificial Intelligence algorithms to determine the movement's angular speed in radians per second (rad/s).

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II) | The evaluation session will be scheduled before of kinematics measurements. The test needs approximately 25-40 minutes to complete.
  The WASI-II is a general intelligence, or IQ test designed to assess specific and overall cognitive capabilities in clinical, educational, and research settings and is individually administered to children, adolescents and adults (ages 6-89). It is a battery of four subtests: Vocabulary (31-item), Block Design (13-item), Similarities (24-item) and Matrix Reasoning (30-item). In addition to assessing general, or Full Scale (range T Scores min 80 - max 320), intelligence, the WASI-II is also designed to provide estimates of Verbal (range T Scores min 40 - max 160) and Performance (range T Scores min 40 - max 160) intelligence consistent with other Wechsler tests. For each scale higher score corresponds to better performance.
Movement Assessment Battery for Children - Second Edition (MABC-2) | The evaluation session will be scheduled before of kinematics measurements. The test needs approximately 20-40 minutes. The checklist needs approximately 10 minutes.
  The MABC-2 identifies and describes impairments in motor performance of children and adolescents 3 through 16 years of age. The MABC-2 consists of 2 components:
  * 24 tests divided into 8 tasks for 3 age groups (3-6; 7-10; 11-16), for 3 areas (Manual dexterity, Aiming and grasping, Balance). There is a total score (TS) and separate scores for the 3 areas. Age-and percentile-adjusted standardized scores are provided for each section of the test and for the TS: TS>67 or a percentile >15th indicates performance in the normal range; 57 <TS> 67 or 6th <percentile >15th defines an "at risk" category with the need for close monitoring; TS ≤56 or percentile ≤5th indicates the presence of a significant motor problem. The test allows to draw a qualitative description of the ways in which the child performs each task;
  * An observation checklist consisting of 43 items divided into 3 sections to be completed by an adult who has the opportunity to observe the child in his daily motor activities.
Behavioral Rating Inventory of Executive Function (BRIEF) | The evaluation session will be scheduled before of kinematics measurements. Questionnaires take 10 minutes to administer.
  The BRIEF-2 is a set of questionnaires for parents and teachers designed to evaluate executive function. The BRIEF-2 now uses 10 clinical scales: Inhibit; Self-Monitor; Shift; Emotional Control; Initiate; Task Completion; Working Memory; Plan/Organize; Task-Monitor; Organization of Materials.
  T scores (min 31 - max >99) and percentile score (min 3 - max >99) are provided for three broad indexes (Behavior Regulation, Emotion Regulation, and Cognitive Regulation) and for the Total Score. Higher score corresponds to better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backstrom A, Johansson AM, Rudolfsson T, Ronnqvist L, von Hofsten C, Rosander K, Domellof E. Motor planning and movement execution during goal-directed sequential manual movements in 6-year-old children with autism spectrum disorder: A kinematic analysis. Res Dev Disabil. 2021 Aug;115:104014. doi: 10.1016/j.ridd.2021.104014. Epub 2021 Jun 24. PMID 34174471
- [Background] Foster NC, Bennett SJ, Causer J, Elliott D, Bird G, Hayes SJ. Getting Off to a Shaky Start: Specificity in Planning and Feedforward Control During Sensorimotor Learning in Autism Spectrum Disorder. Autism Res. 2020 Mar;13(3):423-435. doi: 10.1002/aur.2214. Epub 2019 Oct 29. PMID 31661192
- [Background] Glazebrook CM, Elliott D, Lyons J. A kinematic analysis of how young adults with and without autism plan and control goal-directed movements. Motor Control. 2006 Jul;10(3):244-64. doi: 10.1123/mcj.10.3.244. PMID 17106133
- [Background] Kaur M, M Srinivasan S, N Bhat A. Comparing motor performance, praxis, coordination, and interpersonal synchrony between children with and without Autism Spectrum Disorder (ASD). Res Dev Disabil. 2018 Jan;72:79-95. doi: 10.1016/j.ridd.2017.10.025. Epub 2017 Nov 6. PMID 29121516
- [Background] Grace N, Johnson BP, Rinehart NJ, Enticott PG. Are Motor Control and Regulation Problems Part of the ASD Motor Profile? A Handwriting Study. Dev Neuropsychol. 2018;43(7):581-594. doi: 10.1080/87565641.2018.1504948. Epub 2018 Aug 20. PMID 30124332
- [Background] Vivanti G, Trembath D, Dissanayake C. Mechanisms of imitation impairment in autism spectrum disorder. J Abnorm Child Psychol. 2014 Nov;42(8):1395-405. doi: 10.1007/s10802-014-9874-9. PMID 24736983
- [Background] Zampella CJ, Wang LAL, Haley M, Hutchinson AG, de Marchena A. Motor Skill Differences in Autism Spectrum Disorder: a Clinically Focused Review. Curr Psychiatry Rep. 2021 Aug 13;23(10):64. doi: 10.1007/s11920-021-01280-6. PMID 34387753